CLINICAL TRIAL: NCT03007797
Title: Women - Influencing Factors and Coverage Rate
Brief Title: Realization of the Recommendation for Influenza Vaccination in Pregnant Women
Status: Completed | Type: Observational
Sponsor: University Hospital, Saarland (Other)
Collaborators: Klinikum Worms (Other)
Responsible Party: Sponsor
Other Study IDs: homwo 01
Record Dates: First submitted 2016-12-07; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Coverage Rate of Vaccination for Influenza
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- vaccination rate- pregnant- influenca
  Interventions: Behavioral: vaccination rate for influenza

INTERVENTIONS:
Behavioral: vaccination rate for influenza

SUMMARY:
Introduction:

In 2010, the vaccination recommendations for pregnant women against seasonal influenza were published by the German Standing Committee on Vaccination (STIKO). This work deals with the immunization coverage and the influencing factors.

Method:

A cross-sectional study was realized at two Level 1 perinatal centers in two German federal states during the influenza saisons 2012/2013 and 2013/2014. Pregnant women were interviewed by using a standardized and pre-tested questionnaire covering their knowledge about the influenza vaccination and other factors influencing the vaccination decision. Furthermore, data from the vaccination card and the pregnancy record booklet have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women older than 18
* vaccination records
* signatetd letter of agreement

Exclusion Criteria:

* younger than 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 236 pregnant women in 2 centers
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Influenza Vaccination rate in Pregnant Women | 02/12- 02/14
  The first aim of the study is check how many pregnant women are following the new german recommendation of influenza vaccination in pregnancy.

SECONDARY OUTCOMES:
influencing factors on the Influenza vaccination rate | 02/12- 02/14
  Second aim is to investigate the factors which are influencing the decission for or against the influenza vaccination in pregnancy.